CLINICAL TRIAL: NCT03201575
Title: REmote Ischemic COnditioning in Septic Shock: The RECO-Sepsis Study
Brief Title: REmote Ischemic COnditioning in Septic Shock
Acronym: RECO-Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0290
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Septic Shock
Keywords: Intensive care; septic shock; multiple organ failure; Ischemia-reperfusion; ischemic conditioning; remote conditioning; SOFA score
MeSH Terms: conditions — Shock, Septic; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic conditioning (Experimental): A brachial cuff is positioned around the arm of the patient. The remote ischemic conditioning consists in alternative inflations and deflations of the brachial cuff.
  Interventions: Device: Remote Ischemic conditioning
- Control group (Other): A brachial cuff is positioned around the arm of the patient. No inflation or deflation is made.
  Interventions: Device: Patients with no remote ischemic conditioning

INTERVENTIONS:
Device: Remote Ischemic conditioning — A brachial cuff is positioned around the arm of the patient. Four cycles of [5 min brachial cuff inflation at 200 mmHg followed by 5 min of cuff deflation] started as soon as possible after randomization. The intervention is repeated at 12 and 24 hours after inclusion.
  Arms: Remote ischemic conditioning
Device: Patients with no remote ischemic conditioning — A brachial cuff is positioned around the arm of the patient and no inflation or deflation is made.
  Arms: Control group

SUMMARY:
Septic shock remains a major public health problem in industrialized countries, with a mortality rate as high as 50%, largely related to multiple organ dysfunction. In addition to dysregulated inflammatory response, the pathophysiology of organ failures in septic shock involves ischemia-reperfusion processes. Remote ischemic conditioning is a therapeutic strategy for protecting organs against the detrimental effects of ischemia-reperfusion injury.

The objective of the present study is to determine whether remote ischemic conditioning can limit the severity of organ failure in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hospitalization in an intensive care unit for less than 24 hours
* Septic shock evolving for less than 12 hours defined as:
* Documented or suspected infection
* Norepinephrine administration to maintain a mean arterial pressure ≥ 65 mmHg after volemia correction
* Lactatemia > 2 mmol/L at least once in the past 12 hours before inclusion
* Written informed consent signed by the patient or by a next of kin or oral consent given by the patient and as soon as permitted by the clinical state written informed consent signed by the patient.

Exclusion Criteria:

* Patient who has expressed the wish not to be resuscitated
* Contraindication of the use of brachial cuff on both arms
* Intercurrent pathology with an expected life expectancy of less than 24 hours
* Cardiac arrest
* Female patients currently pregnant or women of childbearing age who are not using contraception
* Previous inclusion in RECO-Sepsis study
* Previous inclusion in another clinical study
* Patients without health coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Average SOFA score (Sequential Organ Failure Assessment) | 96 hours.
  The SOFA score ranges from 0 to 24 (higher scores indicate more severe organ failure), with 0 to 4 points assigned for each of 6 organ dysfunctions (ie, central nervous system, cardiovascular, respiratory, renal, coagulation, and liver).

SECONDARY OUTCOMES:
Average SOFA score without the neurologic sub-score. | 96 hours.
  The SOFA score without the neurologic subscore ranges from 0 to 20 (higher scores indicate more severe organ failure), with 0 to 4 points assigned for each of 5 organ dysfunctions (ie, cardiovascular, respiratory, renal, coagulation, and liver).
SOFA score. | 24 hours
SOFA score. | 48 hours
SOFA score. | 72 hours
SOFA score. | 96 hours
Variations of SOFA score (delta-SOFA) | 24 hours
SOFA sub-scores for each organs | 48 hours
SOFA sub-scores for each organs | 72 hours
SOFA sub-scores for each organs | 96 hours
Survival without organ support | Day 28
Intensive care unit (ICU) length of stay. | Day 90
Hospital length of stay | Day 90
All-cause mortality | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Martin COUR, Principal Investigator — Hospices Civils de Lyon
Locations (6):
- France (6):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Hôpital Edouard Herriot, Lyon
  - CHU de Montpellier, Montpellier
  - CH de Roanne, Roanne
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cour M, Buisson M, Klouche K, Bouzgarrou R, Schwebel C, Quenot JP, Zeni F, Beuret P, Ovize M, Argaud L. Remote ischemic conditioning in septic shock (RECO-Sepsis): study protocol for a randomized controlled trial. Trials. 2019 May 22;20(1):281. doi: 10.1186/s13063-019-3406-4. PMID 31118101
- [Result] Cour M, Klouche K, Souweine B, Quenot JP, Schwebel C, Perinel S, Amaz C, Buisson M, Ovize M, Mewton N, Argaud L; RECO-Sepsis Trial Investigators. Remote ischemic conditioning in septic shock: the RECO-Sepsis randomized clinical trial. Intensive Care Med. 2022 Nov;48(11):1563-1572. doi: 10.1007/s00134-022-06872-1. Epub 2022 Sep 14. PMID 36100725